CLINICAL TRIAL: NCT04925661
Title: Phase Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HEC53856 Capsules in Patients With Non-dialysis Renal Anemia
Brief Title: HEC53856 Phase Ib Study in Patients With Non-dialysis Renal Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Collaborators: Nicoya Therapeutics (Shanghai) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC53856-RAD-102
Record Dates: First submitted 2021-05-30; First posted 2021-06-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2023-04

CONDITIONS: Chronic Kidney Diseases; Renal Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — roxadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The positive drug is Masking and the placebo-controlled is open.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HEC53856 (Experimental): Drug: HEC53856 TIW dosing, capsule There will be a total of 3 dose cohorts: 100mg, 150mg, 200 mg
  Interventions: Drug: HEC53856
- Roxadustat (Active Comparator): Drug: roxadustat TIW dosing There will be only one cohort: 70mg
  Interventions: Drug: Roxadustat
- Placebo (Placebo Comparator): Drug: placebo TIW dosing, capsule There will be a total of 3 dose cohorts: 100mg, 150mg, 200 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HEC53856 — Either dose of HEC53856 will be administered after fasting .
  Arms: HEC53856
Drug: Roxadustat — Roxadustat will be administered after fasting .
  Arms: Roxadustat
Drug: Placebo — Either dose of placebo will be administered after fasting .
  Arms: Placebo

SUMMARY:
To evaluate the safety, tolerability , pharmacokinetics and Preliminary Efficacy of HEC53856 Capsules in Patients With Non-dialysis Renal Anemia.

DETAILED DESCRIPTION:
This is a MultiCenter, Randomized, Blinded, Active Drug and Placebo-controlled, Dose-escalated Phase Ib Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HEC53856 Capsules in Patients With Non-dialysis Renal Anemia. Each part participants will be randomly administrated for HEC53856 or placebo or roxadustat.

The study consisted of three study periods as follows:

Screening period: up to 2 weeks； Treatment period: 8 weeks； Post-Treatment Follow-Up period: 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who agree to participate in this clinical trial and sign an informed consent form;
2. Age 18~65 years old; Weight 40~90Kg, including critical value;
3. Glomerular filtration rate (eGFR) calculated by CKD-EPI formula 15mL/min/1.73 m^2 < or = eGFR < 60 mL/min/1.73 m^2 diagnosed chronic kidney disease patients who have not received dialysis;
4. The hemoglobin values obtained during the last two screening periods at least 6 days apart must be > or = 8.0 g/dL and <10 g/dL.

Exclusion Criteria:

1. Existence of diseases or conditions other than nephropathy that may cause anemia, including but not limited to 1) blood system diseases, such as thalassemia, aplastic anemia, hemolytic anemia, multiple myeloma, myelodysplastic syndrome, etc.; 2) may affect red blood cells The resulting autoimmune diseases, such as systemic lupus erythematosus, rheumatoid arthritis, etc.; 3) Bleeding diseases, such as gastrointestinal bleeding, obstetrics and gynecology bleeding diseases, etc.; 4) Elective surgery expected during the study period;
2. Drugs used to treat anemia within 8 weeks before the first administration, including but not limited to erythropoiesis stimulators (ESAs) and their derivatives, hypoxia inducible factor prolyl hydroxylase inhibitors (HIF-PHI), androgens And anabolic hormone drugs, intravenous iron, Chinese patent medicine, Chinese herbal medicine, etc. (Can accept patients who have used a fixed dose of oral iron within 4 weeks before screening, and continue to take it during the screening period and the first 4 weeks after starting to take the test drug The fixed dose remains unchanged.);
3. Those who have received blood transfusion within 3 months before the first administration;
4. Folic acid <6.8nmol/L (3ng/ml) and (or) VitB12<74pmol/L (100ng/ml) during the screening period;
5. Clinically significant chronic liver and gallbladder disease, or obvious abnormal liver function: ALT>3×ULN and/or AST>3×ULN, or total bilirubin>1.5×ULN;
6. Serum albumin <3 g/dL;
7. The mean systolic blood pressure > or = 160 mmHg and/or the diastolic blood pressure > or = 100 mmHg of the two blood pressure measurements at least one hour apart during the screening period;
8. Suffering from uncontrollable or symptomatic secondary hyperparathyroidism, plasma iPTH > 500pg/ml;
9. A history of acute or chronic pancreatitis, or acute or chronic pancreatitis at the time of screening, or blood amylase > or = 3×ULN;
10. History of malignant tumors within 5 years (except for cured skin basal cell carcinoma and cervical carcinoma in situ), or current assessment of potential malignant tumors;
11. Patients with acute coronary syndrome, stroke ( except for lacunar infarction )or thromboembolic diseases (such as deep vein thrombosis or pulmonary embolism) occurred in the 6 months before screening;
12. New York Society of Cardiology, grade III or IV congestive heart failure, or severe arrhythmia, including but not limited to atrial fibrillation, III degree atrioventricular block, etc.;
13. AIDS antibody, Treponema pallidum antibody, hepatitis B surface antigen or hepatitis C antibody positive for any of them;
14. People with a history of severe allergic disease or drug allergy, or those who are allergic to experimental drugs or their excipients;
15. Patients with clinically severe infections who are receiving systemic antibiotic treatment;
16. Those who have started dialysis or plan to start dialysis treatment within 6 months;
17. Anyone who has participated in or plans to participate in organ transplantation within 6 months;
18. Patients with hemoglobinosis, polycystic kidney disease, or no kidney;
19. Women during pregnancy or lactation, or fertile men and women who refuse to take effective contraceptive measures voluntarily from the beginning of screening to 4 weeks after the administration of the last trial drug;
20. Participated in other clinical trials within 3 months before screening (Definition of participation: accepted trial drug or instrument);
21. The investigator believes that there are other factors that are not suitable for participating in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Through study completion, an average of 12 weeks.
  To assess the safety and tolerability of therapy by incidence of treatment-emergent adverse events after multiple doses of HEC53856 capsule

SECONDARY OUTCOMES:
AUC0-t | Day 1(Dosing) until Day 55 after single and multiple drug dosing.
  Area under the concentration versus time curve (AUC) from time zero to the time of the last quantifiable concentration
Cmax | Day 1(Dosing) until Day 55 after single and multiple drug dosing.
  Maximum observed plasma concentration
Tmax | Day 1(Dosing) until Day 55 after single and multiple drug dosing.
  Time of the maximum observed plasma concentration
T½ | Day 1(Dosing) until Day 55 after single and multiple drug dosing.
  Apparent terminal elimination half-life
Vz/F | Day 1(Dosing) until Day 55 after single and multiple drug dosing.
  Apparent volume of distribution
Changes in mean hemoglobin | week 10
  Changes in mean hemoglobin (Hb) relative to baseline during weeks 8 and 10.
Hemoglobin response | week 10
  Percentage of subjects who met the hemoglobin response after dosing
E-AUC0-t | Day 1(Dosing) until Day 55 after single and multiple drug dosing.
  Area under the EPO concentration versus time curve (AUC) from time zero to the time of the last quantifiable concentration
Emax | Day 1(Dosing) until Day 55 after single and multiple drug dosing.
  Maximum observed EPO concentration
E-Tmax | Day 1(Dosing) until Day 55 after single and multiple drug dosing.
  Time of the maximum observed EPO concentration
Serum lipid | Up to Day 55
  Changes in Serum lipid relative to baseline at weeks 8.
Indicators of iron | Up to Day 55
  Changes in the Indicators of iron relative to baseline at weeks 8.
High-sensitivity C-reactive protein | Up to Day 55
  Changes in the High-sensitivity C-reactive protein relative to baseline at weeks 8.
Reticulocytes | Up to Day 85
  Changes in the mean Reticulocytes relative to baseline after doses.
VEGF | Up to Day 55
  Changes in the VEGF relative to baseline after doses.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - The sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Zhejiang Provincal People's Hospital, Hangzhou
  - The People's Hospital of Guangxi Zhuang Autonmous Region, Nanning
  - Huashan Hospital, Shanghai
  - Ruijin Hospital, Shanghai
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen